CLINICAL TRIAL: NCT02692625
Title: Consumption Effect of Probiotic Products on Salivary Cariogenic Bacterial Counts in Preschool Children.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Najlaa Alamoudi, Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KAUFD
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A (test group): This group consist of 80 children receiving the probiotic lozenges.
  The Probiotic lozenges used in the trial is a non-commercial product provided by BioGaia AB, Lund, Sweden. The Probiotic lozenges consist of a minimum of 200 million live L. reuteri (L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289 (L. reuteri Prodentis®). The probiotic lozenge is used twice daily for two months.
  Interventions: Dietary Supplement: (L. reuteri Prodentis®).
- Group B (Placebo Comparator): Group B (control group): This group consist of 80 children receiving the placebo lozenges.
  The placebo lozenges used in the trial is non-commercial product provided by BioGaia AB, Lund, Sweden.The placebo lozenges is used twice daily for two months.
  Interventions: Dietary Supplement: Placebo lozenges

INTERVENTIONS:
Dietary Supplement: (L. reuteri Prodentis®). — The Test group is instructed to consume Probiotic lozenges for two months. The counts of salivary mutans streptococci and lactobacilli were evaluated using the CRT test at baseline, one-month, and two- months, from the beginning of the trial for every participating child.
  Arms: Group A
Dietary Supplement: Placebo lozenges — The control group is instructed to consume placebo lozenges for two months. The counts of salivary mutans streptococci and lactobacilli were evaluated using the CRT test at baseline, one-month, and two- months, from the beginning of the trial for every
  Arms: Group B

SUMMARY:
The purpose of this study is to evaluate the efficacy of probiotic products on caries-associated salivary bacterial counts (Streptococcus mutans and Lactobacillus) and its effect on dental plaque accumulation in a group of preschool children in Saudi Arabia.

DETAILED DESCRIPTION:
Among the dental conditions that are most common among the children is dental caries. This condition can afflict an individual in the course of their entire life. However, it is possible to develop prevention mechanisms especially during childhood (1). Dental caries can be defined as the damage of a specific susceptible part of the enamel through acids that are produced by bacteria as they ferment carbohydrates that have been trapped within the teeth (2). A number of endogenous bacteria are known of producing acidic by-products, which ends up destroying the tooth. Some of the notorious bacteria are Streptococci mutans, Lactobacillus spp. and Streptococcus sobrinus. Release of acids through fermentation cause a fall in pH causing decalcifying of the structure of enamel, thereby causing irreversible damage in form of caries (3, 4). Recent research studies have indicated that the use of probiotics provides a future prevention solution against caries. The use of probiotic therapy is based on the fact that the oral cavity has a specific ecosystem of bacteria comprising of normal flora and pathogenic bacteria, which live together. Probiotic therapy seeks to balance this oral ecosystem so as to ensure that harmful bacteria are eliminated. An imbalance in oral ecosystem can cause dental caries, for example, streptococcus mutans, which form part of the normal oral flora can result to decalcification of the enamel if their numbers rise beyond normal. Probiotic is a derivative of Greek work, which means "for life," it was first used in 1965 by Lilly and Stillwell and was found to be a contrast of the antibiotic (5). WHO/FAO (2002) defines probiotics as living organisms that have health benefits to the host when administered in the desirable amounts. In a number of studies on probiotics, the focus has been on reducing the number of mutans streptococci. The most widely used probiotic strains are Lactobacillus and Bifidobacterium. Irrespective of the strain or product used, various studies point to reduced number of mutans streptococci in saliva, an effect that is widely varied with the study groups being small (6,7,8,9) and conducted over a short period (6,7,8,9,10). Based on these findings, the efficacy of probiotic chewable tablets in prevention of caries require further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children having no history of any systemic conation, having full set of primary dentition, having high counts of salivary mutants streptococci ( ≥ 105 CFU ), dft score ≥ 3, with no history of recent antibiotics administration (At least one month prior to the intervention) .

Exclusion Criteria:

* Disapproved consent, medically compromised children, children using topical fluoride within the 4 weeks prior to baseline except the fluoride in the toothpaste, and children using xylitol chewing gums.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The salivary mutans streptococci and lactobacilli counts | 2 months

SECONDARY OUTCOMES:
Dental plaque accumulation. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Najlaa M Alamoudi, BDS, MS, DS, Principal Investigator — King Abdulaziz University
Locations (1):
- King abulaziz University, Dental University Hospital, Jeddah, P.O Box 80209, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kidd EA, Fejerskov O. What constitutes dental caries? Histopathology of carious enamel and dentin related to the action of cariogenic biofilms. J Dent Res. 2004;83 Spec No C:C35-8. doi: 10.1177/154405910408301s07. PMID 15286119
- [Result] Featherstone JD. The continuum of dental caries--evidence for a dynamic disease process. J Dent Res. 2004;83 Spec No C:C39-42. doi: 10.1177/154405910408301s08. PMID 15286120
- [Result] LILLY DM, STILLWELL RH. PROBIOTICS: GROWTH-PROMOTING FACTORS PRODUCED BY MICROORGANISMS. Science. 1965 Feb 12;147(3659):747-8. doi: 10.1126/science.147.3659.747. PMID 14242024
- [Result] Aminabadi NA, Erfanparast L, Ebrahimi A, Oskouei SG. Effect of chlorhexidine pretreatment on the stability of salivary lactobacilli probiotic in six- to twelve-year-old children: a randomized controlled trial. Caries Res. 2011;45(2):148-54. doi: 10.1159/000325741. Epub 2011 Mar 31. PMID 21454978
- [Result] Cildir SK, Sandalli N, Nazli S, Alp F, Caglar E. A novel delivery system of probiotic drop and its effect on dental caries risk factors in cleft lip/palate children. Cleft Palate Craniofac J. 2012 May;49(3):369-72. doi: 10.1597/10-035. Epub 2011 Feb 10. PMID 21309653
- [Result] Sudhir R, Praveen P, Anantharaj A, Venkataraghavan K. Assessment of the effect of probiotic curd consumption on salivary pH and streptococcus mutans counts. Niger Med J. 2012 Jul;53(3):135-9. doi: 10.4103/0300-1652.104382. PMID 23293413
- [Result] Juneja A, Kakade A. Evaluating the effect of probiotic containing milk on salivary mutans streptococci levels. J Clin Pediatr Dent. 2012 Fall;37(1):9-14. doi: 10.17796/jcpd.37.1.tq91178m7w876644. PMID 23342560